CLINICAL TRIAL: NCT01659931
Title: A Single Dose, Two-Period, Two-Treatment, Two-Way Crossover Bioequivalence Study of Montelukast Sodium 10 mg Tablets Under Fasted Conditions
Brief Title: Bioequivalency Study of Montelukast 10 mg Tablets Under Fasted Conditions
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Sponsor
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MONT-T10-PVFS-1
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Montelukast (Active Comparator): 10 mg Tablet
  Interventions: Drug: Montelukast
- Singulair (Active Comparator): 10 mg Tablet
  Interventions: Drug: Singulair

INTERVENTIONS:
Drug: Montelukast — 10 mg Tablet
  Other Names: Singulair
  Arms: Montelukast
Drug: Singulair — 10 mg Tablet
  Other Names: Montelukast
  Arms: Singulair

SUMMARY:
The objective of this study was to prove the bioequivalence of Montelukast Tablet under fasted conditions

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to montelukast or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2008-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
bioequivalence determined by statistical comparison Cmax | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Alan K Copa, PharmD, Principal Investigator — PRACS Institute, Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States